CLINICAL TRIAL: NCT03492593
Title: Métabolismes Des caroténoïdes Dans la lumière du Tube Digestif de l'Homme Sain
Brief Title: Lycopene and Beta-carotene Metabolism in the Digestive Tract of Healthy Men
Acronym: CarotenoiDig
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Aix Marseille Université (Other); Hôpital de la Conception (Unknown)
Responsible Party: Principal Investigator, Patrick Borel, Principal Investigator, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013-A01398-37; 2013-A01398-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Digestion Chambers; Stability and Metabolism of Carotenoids and Vitamin E
Keywords: carotenoids; vitamin E; digestion; stability; metabolism
MeSH Terms: interventions — Lycopene; beta Carotene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- lycopene (Experimental): A dose of lycopene (20 mg) is provided as part of an emulsified liquid meal (with or without 160 mg powdered ferrous sulfate). Samples from the upper digestive tract (gastric or duodenal) are aspirated over 4 hours, and blood collected over 7 hours. Blood plasma and chylomicron fractions isolated. The subject returns for 3 additional visits with 2 weeks between each visit. The same protocol is followed, with the subject receiving all combinations of meal (w/ and w/o iron) and upper digestive tract sampling (gastric or duodenal)
  Interventions: Other: lycopene
- 13C beta-carotene (Experimental): A dose of 13C beta-carotene (20 mg) is provided as part of an emulsified liquid meal. Samples from the upper digestive tract (gastric or duodenal) are aspirated over 5 hours, blood collected over 7 hours, and urine collected over 7 hours. Blood plasma and chylomicron fractions isolated. The subject returns for 1 additional visit with a minimum of 4 weeks between each visit. The same protocol is followed, with sampling taken from the remaining upper digestive tract compartment (gastric or duodenal)
  Interventions: Other: beta-carotene
- control (Placebo Comparator): The same procedure is followed (as detailed in the experimental arms) but the subject receives an emulsified liquid meal without carotenoids or vitamin E.
  Interventions: Other: control

INTERVENTIONS:
Other: lycopene — A tomato oleoresin containing lycopene
  Arms: lycopene
Other: beta-carotene — 13C beta-carotene
  Arms: 13C beta-carotene
Other: control — emulsified liquid meal alone
  Arms: control

SUMMARY:
Consumption of foods containing carotenoids, as well as vitamin E, have been associated with lower risk of developing a number of chronic diseases. While the parent compounds have largely been assumed to exert protective antioxidant effects, more recent work has suggested that metabolites may be bioactive. Very little attention has been given to the metabolism of these compounds during the digestive process. Our primary aim is to conduct a postprandial feeding study in healthy men to determine the stability of carotenoids and vitamin E during digestion, and to identify the primary metabolites produced in various compartments of the upper gastrointestinal tract and blood during digestion. Targeted metabolites will be identified and quantitated using high-performance liquid chromatography-tandem mass spectrometry methods previously developed. In addition, a non-targeted metabolomics approach will be used to identify non-predicted metabolites in the samples. A better understanding of carotenoid and vitamin E stability and metabolism during digestion will provide greater insight into how these compounds may confer protection against chronic disease.

DETAILED DESCRIPTION:
Consumption of foods containing the carotenoids lutein, lycopene, beta-carotene, as well as vitamin E, have been associated with lower risk of developing chronic diseases including cardiovascular disease, cancer, age related macular degeneration, and cognitive decline. While the parent compounds have largely been assumed to exert protective antioxidant effects, more recent work has suggested that metabolites may be bioactive. Very little attention has been given to the metabolism of these compounds during the digestive process. Our primariy aim is to conduct a postprandial feeding study in healthy men to determine the stability of carotenoids and vitamin E during digestion, and to identify the primary metabolites produced in the upper gastrointestinal tract during digestion. Subjects will be fed a meal containing either lutein,lycopene, deuterated beta-carotene, or deuterated vitamin E. Gastric and duodenal samples will be taken 5 hours post-meal consumption, while blood plasma and chylomicron fractions will be taken over 7 hours post-meal consumption. Targeted metabolites will be identified and quantitated using high-performance liquid chromatography-tandem mass spectrometry methods previously developed. In addition, a non-targeted metabolomics approach will be used to identify non-predicted metabolites in a subset of collected samples. Overall, this research will provide very original insight about carotenoid and vitamin E metabolites produced during the digestive process and their absorption by the human body. This information is essential to understand how these compounds may confer protection against chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18-29.9
* Cholesterol < 2.2 g/L
* Triglycerides < 1.5 g/L
* Blood sugar </= 1.1 g/L
* Hemoglobin > 13 g/dL
* Test negative for hepatitis B, C, and HIV

Exclusion Criteria:

* Hepatitis B and C
* HIV
* Blood donation or blood sampling less than 2 months prior to the first daylong study day
* Craniofacial trauma
* Smokers
* Regular consumption of vitamins or supplements rich in carotenoids or vitamin E in the past 3 months
* Alcohol consumption > 140 g per week (equivalent to 14 glasses of wine, 14 glasses of beer (25 mL), or 14 shots of liquor).
* Past or present eating disorder (anorexia, bulimia, etc.)
* Food allergies to components of the liquid test meal
* Medical treatment or surgical intervention affecting the digestive tract or function of the digestive tract
* Metabolic disorders (disorder of the liver or pancreas, diabetes, hemochromatosis, gastro-intenstinal disorders with the exception of appendicitis)
* Use of certain medications (those which regulate intestinal transit, those which reduce blood lipids and cholesterol, those which interact with bile salts)
* All medical indications which fall within the context of exclusion criteria as determined by the supervising physician of the study
* Intense physical activity > 4 1/2 hours per week
* Participation in another clinical study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Lycopene Metabolites | 7 hours
beta-carotene metabolites | 7 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Borel, PhD, Principal Investigator — INRA/INSERM/Université Aix-Marseille; Catherine Caris-Veyrat, Study Director — INRA/Université d'Avignon
Locations (1):
- Centre d'Investigation Clinique de la Hôpital Conception, Marseille, France

REFERENCES:
- [Derived] Kopec RE, Caris-Veyrat C, Nowicki M, Gleize B, Carail M, Borel P. Production of asymmetric oxidative metabolites of [13C]-beta-carotene during digestion in the gastrointestinal lumen of healthy men. Am J Clin Nutr. 2018 Oct 1;108(4):803-813. doi: 10.1093/ajcn/nqy183. PMID 30256893